CLINICAL TRIAL: NCT01730937
Title: Randomized Phase III Study of Sorafenib Versus Stereotactic Body Radiation Therapy Followed by Sorafenib in Hepatocellular Carcinoma
Brief Title: Sorafenib Tosylate With or Without Stereotactic Body Radiation Therapy in Treating Patients With Liver Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RTOG-1112; NCI-2012-02057 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U10CA021661 (NIH)
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Results first posted 2023-07-03 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-09

CONDITIONS: Adult Primary Hepatocellular Carcinoma; Advanced Adult Primary Liver Cancer; Recurrent Adult Primary Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; Radiosurgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib Alone (Active Comparator): 400 mg sorafenib twice a day for 28-day cycle. Continue up to 5 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Sorafenib
- SBRT followed by Sorafenib (Experimental): 27.5 Gy to 50 Gy stereotactic body radiation therapy (SBRT) in 5 fractions 24-72 hours apart over 5-15 days followed within 1-5 days by one cycle of 200 mg sorafenib twice a day. Starting with second cycle, if tolerable, increase to 400 mg sorafenib twice a day. Continue up to 5 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Sorafenib; Radiation: stereotactic body radiation therapy

INTERVENTIONS:
Drug: Sorafenib — By mouth (PO)
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN; Sorafenib Tosylate
Radiation: stereotactic body radiation therapy — Intensity-modulated radiation therapy (IMRT), stereotactic body radiation therapy (SBRT), and proton therapy are allowed.
  Other Names: SBRT; stereotactic radiation therapy; stereotactic radiotherapy; stereotactic ablative body radiation therapy,; stereotactic ablative radiotherapy; SABR
  Arms: SBRT followed by Sorafenib

SUMMARY:
This randomized phase III trial studies sorafenib tosylate and stereotactic body radiation therapy to see how well they work compared to sorafenib tosylate alone in treating patients with liver cancer. Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Stereotactic body radiation therapy may be able to send the radiation dose directly to the tumor and cause less damage to normal tissue. Giving sorafenib tosylate together with stereotactic body radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if stereotactic body radiation therapy (SBRT) improves overall survival in hepatocellular carcinoma (HCC) patients treated with sorafenib (sorafenib tosylate).

SECONDARY OBJECTIVES:

I. To determine the difference in time to progression (TTP) and progression-free survival (PFS) in HCC patients treated with sorafenib compared to SBRT followed by sorafenib.

II. To measure differences in toxicity in HCC patients treated with sorafenib versus SBRT followed by sorafenib.

III. To measure vascular thrombosis response post sorafenib versus SBRT followed by sorafenib.

IV. To measure differences in health related quality of life (QOL) and quality-adjusted survival in HCC patients treated with sorafenib compared to SBRT followed by sorafenib.

V. Collection of biospecimens for future correlative studies to investigate differences in potential biomarkers in patients treated with sorafenib versus SBRT followed by sorafenib.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of HCC by at least one criterion listed below within 360 days prior to study entry:

  * Pathologically (histologically or cytologically) proven diagnosis of HCC,(biopsies are recommended, and are to be submitted for research evaluation if patients consent)
  * At least one solid liver lesion or vascular tumor thrombosis (involving portal vein, inferior vena cava (IVC) and/or hepatic vein) > 1 cm with arterial enhancement and delayed washout on multi-phasic computerized tomography (CT) or magnetic resonance imaging (MRI) in the setting of cirrhosis or chronic hepatitis B or C without cirrhosis.
  * For patients whose CURRENT disease is vascular only: enhancing vascular thrombosis (involving portal vein, IVC and/or hepatic vein) demonstrating early arterial enhancement and delayed washout on multi-phasic CT or MRI in a patient with known HCC (diagnosed previously <720 days) using the above criteria.
* Measureable hepatic disease and/or presence of vascular tumor thrombosis (involving portal vein, IVC and/or hepatic vein) which may not be measureable as per Response Evaluation Criteria in Solid Tumors (RECIST) on liver CT or MRI, within 28 days of registration
* Appropriate for protocol entry based upon the following minimum diagnostic workup:

  * History/physical examination including examination for encephalopathy, ascites, weight, height, and blood pressure within 14 days prior to study entry
  * Assessment by radiation oncologist and medical oncologist or hepatologist who specializes in treatment of HCC within 28 days prior to study entry
  * Pre-randomization Scan (REQUIRED for All Patients): Within 28 days prior to study entry, multiphasic liver CT or multiphasic liver MR scan.
  * Within 28 days prior to study entry CT chest with CT or MR abdomen and CT or MR pelvis, or positron emission tomography (PET) CT chest/abdomen/pelvis.
* Zubrod performance status 0-2 within 28 days prior to study entry
* All blood work obtained within 14 days prior to study entry with adequate organ marrow function defined as follows:

  * Absolute neutrophil count (ANC) >= 1,500 cells/mm^3
  * Platelets >= 60,000 cells/mm^3
  * Hemoglobin >= 8.0 g/dl (note: the use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 8.0 g/dl is acceptable)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 6 times upper limit of normal (ULN)
  * Serum creatinine =< 2 x ULN or creatinine clearance >= 60 mL/min
* Barcelona Clinic Liver Cancer (BCLC) stage: intermediate (B) or advanced (C) within 28 days prior to study entry
* Child-Pugh score A within 14 days prior to study entry
* Women of childbearing potential and male participants must agree to practice adequate contraception while on study and for at least 6 months following the last dose of radiation therapy (RT) and for at least 28 days following the last dose of sorafenib (whichever is later)
* Unsuitable for resection or transplant or radiofrequency ablation (RFA)
* Unsuitable for or refractory to transarterial hepatic chemo-embolization (TACE) or drug eluting beads (DEB) for any of the following reasons, as described by Raoul et al (2011):

  * Technical contraindications: arteriovenous fistula, including, surgical portosystemic shunt or spontaneous portosystemic shunt
  * Severe reduction in portal vein flow: due to tumor portal vein, IVC or atrial invasion or bland portal vein occlusion
  * Medical contraindications including congestive heart failure, angina, severe peripheral vascular disease
  * Presence of extrahepatic disease
  * No response post TACE (or DEB) or progressive HCC despite TACE; prior TACE or DEB is allowed but must be > 28 days from study entry
  * Serious toxicity following prior TACE (or DEB); prior TACE or DEB must be > 28 days from study entry
  * Other medical comorbidities making TACE (or DEB) unsafe and/or risky (e.g. combination of relative contraindications including age > 80 years, tumor > 10 cm, > 50% replacement of the liver by HCC, extensive multinodular bilobar HCC, biliary drainage)
* Patients treated with prior surgery are eligible for this study if they otherwise meet eligibility criteria
* Patient must be able to provide study-specific informed consent prior to study entry

Exclusion Criteria:

* Prior invasive malignancy (except non-melanomatous skin cancer and T1 renal cell carcinoma) unless disease free for a minimum of 2 years (note that carcinoma in situ of the breast, oral cavity, or cervix are all permissible)
* Prior sorafenib use > 60 days and/or grade 3 or 4 sorafenib related toxicity. Note that prior chemotherapy for HCC or a different cancer is allowable
* Prior radiotherapy to the region of the liver that would result in overlap of radiation therapy fields
* Prior selective internal radiotherapy/hepatic arterial yttrium therapy, at any time
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months PRIOR TO registration
  * Transmural myocardial infarction within the last 6 months prior to study entry
  * Unstable ventricular arrhythmia within the last 6 months prior to study entry
  * Acute bacterial or fungal infection requiring intravenous antibiotics within 28 days prior to study entry
  * Hepatic insufficiency resulting in clinical jaundice, encephalopathy and/or variceal bleed within 28 days prior to study entry
  * Bleeding within 28 days prior to study entry due to any cause, requiring transfusion
  * Thrombolytic therapy within 28 days prior to study entry. Subcutaneous heparin is permitted.
  * Known bleeding or clotting disorder
  * Uncontrolled psychotic disorder
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic
* Maximal diameter of any one hepatocellular carcinoma > 15 cm
* Total sum of maximum diameters of each definite parenchymal hepatocellular carcinoma within the liver or maximum diameter of a single conglomerate HCC > 20 cm
* More than 5 discrete intrahepatic parenchymal foci of HCC
* Direct tumor extension into the stomach, duodenum, small bowel or large bowel
* Measureable common or main branch biliary duct involvement with HCC
* Extrahepatic metastases or malignant nodes (that enhance with typical features of HCC) > 3.0 cm, in sum of maximal diameters (e.g. presence of one 3.4 cm metastatic lymph node or two 2 cm lung lesions); note that benign non-enhancing periportal lymphadenopathy is not unusual in the presence of hepatitis and is permitted, even if the sum of enlarged nodes is > 2.0 cm
* Prior liver transplant
* HIV positive with CD4 (T-cell count) count < (350) cells/microliter. Note that patients who are HIV positive are eligible, provided they are under treatment with highly active antiretroviral therapy (HAART) and have a CD4 count ≥ (350) cells/microliter, and no known detectable viral load, at the time of study entry. Note also that HIV testing is not required for eligibility for this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2025-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Dawson, Principal Investigator — Radiation Therapy Oncology Group
Locations (51):
- United States (41):
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - University of Colorado Hospital, Aurora, Colorado
  - Saint Vincent's Medical Center, Bridgeport, Connecticut
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Queen's Medical Center, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Hunter Holmes McGuire Veterans Administration Medical Center, Richmond, Virginia
  - ProCure Proton Therapy Center-Seattle, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia
- Canada (7):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
- Pamela Youde Nethersole Eastern Hospital, Chai Wan, Hong Kong
- Samsung Medical Center, Seoul, Korea, South Korea

REFERENCES:
- [Derived] Dawson LA, Winter KA, Knox JJ, Zhu AX, Krishnan S, Guha C, Kachnic LA, Gillin MT, Hong TS, Craig TD, Williams TM, Hosni A, Chen E, Noonan AM, Koay EJ, Sinha R, Lock MI, Ohri N, Dorth JA, Delouya G, Swaminath A, Moughan J, Crane CH. Stereotactic Body Radiotherapy vs Sorafenib Alone in Hepatocellular Carcinoma: The NRG Oncology/RTOG 1112 Phase 3 Randomized Clinical Trial. JAMA Oncol. 2025 Feb 1;11(2):136-144. doi: 10.1001/jamaoncol.2024.5403. PMID 39699905

RESULTS

PARTICIPANT FLOW:
Groups:
- Sorafenib Alone: 400 mg sorafenib by mouth twice a day for 28-day cycle. Continue up to 5 years in the absence of disease progression or unacceptable toxicity.
- SBRT Followed by Sorafenib: 27.5 Gy to 50 Gy stereotactic body radiation therapy (SBRT) in 5 fractions 24-72 hours apart over 5-15 days followed within 1-5 days by one cycle of 200 mg sorafenib by mouth twice a day. Starting with second cycle, if tolerable, increase to 400 mg sorafenib by mouth twice a day. Continue up to 5 years in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Sorafenib Alone | SBRT Followed by Sorafenib
Started | 97 | 96
Eligible Population | 92 | 85
Adverse Event Population (Eligible, started treatment, and were assessed for adverse events.) | 88 | 83
Quality of Life Population (Eligible with consent for quality of life study component) | 46 | 37
Completed (Participants contributing data to results are considered to have completed the study.) | 92 | 85
Not Completed | 5 | 11
Not completed — Protocol Violation | 5 | 11

BASELINE CHARACTERISTICS:
Population: Eligible participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib Alone | SBRT Followed by Sorafenib | Total
Number analyzed (Participants) | 92 | 85 | 177
Age, Continuous [Median (Full Range); unit: years] | 67 [27 to 84] | 66 [49 to 83] | 66 [27 to 84]
Age, Customized [Count of Participants; unit: Participants]
  ≤ 49 years | 3 | 1 | 4
  50 - 59 years | 15 | 20 | 35
  60 - 69 years | 39 | 42 | 81
  70 - 79 years | 26 | 18 | 44
  ≥ 80 years | 9 | 4 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 17 | 27
  Male | 82 | 68 | 150
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 8
  Not Hispanic or Latino | 54 | 47 | 101
  Unknown or Not Reported | 32 | 36 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 23 | 18 | 41
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 5 | 3 | 8
  White | 58 | 59 | 117
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 9
Zubrod performance status [Count of Participants; unit: Participants] — 0 - Asymptomatic; 1 - Symptomatic but completely ambulatory; 2 - Symptomatic, <50% in bed during the day; 3 - Symptomatic, >50% in bed, but not bedbound; 4 - Bedbound; 5 - Death
  Participants
    0 | 41 | 47 | 88
    1 | 44 | 33 | 77
    2 | 7 | 5 | 12
T Stage [Count of Participants; unit: Participants] — Tumor stage per the American Joint Committee on Cancer (AJCC) 7th ed. refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. T's may be further divided to provide more detail, such as T3a and T3b.
  Participants
    T1 | 9 | 6 | 15
    T2 | 17 | 19 | 36
    T3a | 12 | 16 | 28
    T3b | 49 | 38 | 87
    T4 | 5 | 6 | 11
N Stage [Count of Participants; unit: Participants] — Regional lymph nodes staging per American Joint Committee on Cancer (AJCC) 7th ed. refers to the number and/or extent of spread of lymph nodes that contain cancer. The higher the number after the N, the greater the involvement of regional lymph nodes. (N0= no cancer in nearby lymph nodes; NX = cannot be measured.)
  Participants
    N0 | 89 | 80 | 169
    N1 | 3 | 4 | 7
    NX | 0 | 1 | 1
M Stage [Count of Participants; unit: Participants] — Metastasis stage per the American Joint Committee on Cancer (AJCC) 7th ed. refers to the spread of the cancer to organs and tissues in other parts of the body. M0 = No distant metastasis; M1 = Distant metastasis; MX = Distant metastasis cannot be assessed.
  Participants
    M0 | 88 | 82 | 170
    M1 | 4 | 3 | 7
Child Pugh Score [Count of Participants; unit: Participants] — Child Pugh Classification uses the following to determine liver function: 1) bilirubin levels; 2) albumin levels; 3) how quickly the blood clots (prothrombin time); 4) if there is fluid in the abdomen (ascites); and 5) if there is encephalopathy (liver disease has affected brain function). Each one of the previous is given a score: 5 (Grade A) and 6 (Grade A) mean the liver is working normally.
  Participants
    5 (Grade A) | 69 | 64 | 133
    6 (Grade A) | 23 | 21 | 44
BCLC Stage [Count of Participants; unit: Participants] — Barcelona Clinic Liver Cancer (BCLC) staging system helps doctors determine the best treatment using 1) the number and size of tumors in the liver, 2) general health status or Zubrod performance status, and 3) liver function using Child-Pugh score. Intermediate(B): many tumors in liver, but overall status is good (Zubrod=0) and liver function is good with Child Pugh A or B. Advanced(C): cancer has spread, Zubrod=1 or 2, but liver function is still good with Child Pugh A or B.
  Participants
    Intermediate (B) | 15 | 17 | 32
    Advanced (C) | 77 | 68 | 145
Hepatocellular carcinoma (HCC) tumor volume / liver volume [Count of Participants; unit: Participants] — The ratio of hepatocellular volume to the liver volume (as a percent).
  Participants
    <10% | 40 | 40 | 80
    10-40% | 42 | 39 | 81
    >40% | 10 | 6 | 16
Hepatitis Status [Count of Participants; unit: Participants] — Hepatitis is a type of liver disease that causes inflammation of the liver, which can be caused by alcohol, injury, autoimmune response, or a reaction to bacteria or virus. Hepatitis B may result in chronic liver disease or liver cancer. Hepatitis C may result in cirrhosis or liver cancer. Other (Hepatitis A) mostly likely will result in no liver damage.
  Participants
    Hepatitis B or B and C | 17 | 16 | 33
    Hepatitis C | 38 | 35 | 73
    Other | 37 | 34 | 71
Enhancing vascular thrombosis [Count of Participants; unit: Participants]
  Yes | 66 | 62 | 128
  No | 26 | 23 | 49
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 90 | 85 | 175
  Other | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: An event for overall survival (OS) is death due to any cause. Survival time is defined as time from randomization to the date of death or last known follow-up (censored). Rates are estimated by the Kaplan-Meier method. Analysis was to occur after 153 deaths were reported.
Time Frame: From randomization to last follow-up: weekly during SBRT, post-SBRT/pre-sorafenib, monthly during sorafenib, and overall, from study entry: every 3 months for 2 years, then every 6 months. Maximum follow-up at time of analysis was 7.6 years.
Population: Eligible participants
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Sorafenib Alone | SBRT Followed by Sorafenib
Number analyzed (Participants) | 92 | 85
months | 12.30 [10.62 to 14.3] | 15.85 [11.42 to 19.15]
Statistical Analysis 1: Comparison: Sorafenib Alone vs SBRT Followed by Sorafenib; Original design: Hypothesized 28% reduction (HR=0.72) with SBRT (corresponds to median OS = 14.5 months). Assuming an exponential distribution and constant hazards, 292 patients were required to reach 238 OS events, with 80% statistical power, a 1-sided α of 0.05. Revised design (see limitations/caveats): For same above hypotheses, at least 155 OS events from 193 randomized patients provided 65% statistical power, with a 1-sided α of 0.05; Test type: Superiority; p = 0.0554, Log Rank; Hazard Ratio (HR) = 0.77, 90% CI 2-sided [0.59 to 1.01] — Reference arm = Sorafenib Alone

2. Secondary Outcome: Time to Progression
Description: Progression (failure) is defined as any of the following events: new tumor thrombosis, progression of hepatocellular carcinoma (HCC) within liver excluding tumor thrombosis status, progression of distant metastases that were present at study entry, new HCC within the liver including tumor thrombosis, and vascular thrombosis events=progression-new enhancing tumor thrombosis/progression-Increase in the volume of enhancing portion of thrombosis. Time to progression was measured from the date of randomization to the date of first failure, death (competing risk), or last follow-up (censored). Progression rates are estimated by the cumulative incidence method. The protocol specifies only that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Two-year estimates are provided as a summary of the distributions.
Time Frame: as for outcome 1
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sorafenib Alone | SBRT Followed by Sorafenib
Number analyzed (Participants) | 92 | 85
percentage of participants | 66.3 [55.3 to 75.3] | 56.4 [44.9 to 66.4]
Statistical Analysis 1: Comparison: Sorafenib Alone vs SBRT Followed by Sorafenib; Test type: Superiority; p = 0.034, Gray's test — Two-sided significance level = 0.05; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.48 to 0.99] — Reference arm = Sorafenib Alone

3. Secondary Outcome: Progression-free Survival
Description: Failure for progression-free survival (PFS) include death, new tumor thrombosis, progression of hepatocellular carcinoma (HCC) within liver excluding tumor thrombosis status, progression of distant Mets that were present at study entry, new HCC within liver including tumor thrombosis, and vascular thrombosis events =progression-new enhancing tumor thrombosis/progression-Increase in the volume of enhancing portion of thrombosis. PFS time is defined as the time from randomization to the date of first failure, date of death, or last known follow-up (censored). PFS rates are estimated by the Kaplan-Meier method. The protocol specifies only that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Two-year estimates are provided as a summary of the distributions.
Time Frame: as for outcome 1
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sorafenib Alone | SBRT Followed by Sorafenib
Number analyzed (Participants) | 92 | 85
percentage of participants | 5.49 [3.42 to 6.28] | 9.22 [7.53 to 11.89]
Statistical Analysis 1: Comparison: Sorafenib Alone vs SBRT Followed by Sorafenib; Test type: Superiority; p = 0.0001, Log Rank — Two-sided significance level=0.05; Hazard Ratio (HR) = 0.55, 95% CI 2-sided [0.40 to 0.75] — Reference arm = Sorafenib Alone

4. Secondary Outcome: Number of Participants by Highest Grade Adverse Event Reported
Description: Common Terminology Criteria for Adverse Events (version 4.0) grades adverse event severity from 1=mild to 5=death. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data.
Time Frame: as for outcome 1
Population: Eligible, started treatment, and were assessed for adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib Alone | SBRT Followed by Sorafenib
Number analyzed (Participants) | 88 | 83
Participants
  Grade 1 | 2 | 1
  Grade 2 | 21 | 20
  Grade 3 | 49 | 51
  Grade 4 | 10 | 9
  Grade 5 | 6 | 2

5. Secondary Outcome: Percentage of Participants With Improvement in the Functional Assessment of Cancer Therapy - Hepatobiliary (FACT-Hep) Total Score 6 Months After the Start of Treatment
Description: The FACT-Hep total score measures quality of life in patients with hepatobiliary cancer. Possible scores range from 0 to 180, with higher scores indicating a better outcome. Improvement in FACT-Hep total score is defined as an increase from the baseline to 6-month score of at least 5 points.
Time Frame: Baseline and 6 months
Population: Eligible participants who consented to the quality of life component and had data at baseline and six months.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sorafenib Alone | SBRT Followed by Sorafenib
Number analyzed (Participants) | 20 | 17
percentage of participants | 10 [2 to 31] | 35 [17 to 59]

6. Secondary Outcome: Best Vascular Thrombosis Response up to the Time of Progressive Disease (if Applicable)
Description: Complete response: Complete resolution of thrombosis, with recanalization of vessel.
  Partial response (PR):
  * Partial recanalization (if prior complete blockage)
  * Unequivocal reduction in the maximal girth
  * Unequivocal reduction in the volume, or elimination, of arterial enhancing portion
  Progressive disease (PD): any unequivocal, unambiguous
  * New enhancing tumor thrombosis
  * Increase in the volume of enhancing portion
  * Unequivocal progression of thrombosis (non-measurable disease), the increase in overall tumor burden (enhancing thrombosis) must be comparable to the increase required for the Response Evaluation Criteria in Solid Tumor 1.1 definition of PD of measurable disease (e.g. ≥ 73% increase in volume, which is similar to 20% increase in diameter, and at least a 5 mm absolute increase).
  Stable disease:
  * No/small changes that do not meet the above criteria for PR or PD
  * Increase in the volume of non-enhancing thrombosis
  * New bland non-enhancing thrombosis
Time Frame: From randomization to last follow-up. Imaging occurs every 3 months for two years then every six months. Maximum follow-up at time of analysis was 7.6 years.
Population: Eligible participants who had vascular thrombosis at study entry
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib Alone | SBRT Followed by Sorafenib
Number analyzed (Participants) | 66 | 62
Participants
  Complete Response | 0 | 2
  Partial Response | 6 | 22
  Stable Disease | 25 | 23
  Progressive Disease | 14 | 4
  Unknown | 21 | 11

7. Secondary Outcome: Quality Adjusted Life Years
Description: Quality adjusted life years is calculated as the weighted sum of the number of years spent in different health states. The weight value is a utility score between 0 (worst health state) and 1 (best health state) derived from the EQ-5D-5L questionnaire, designed to describe and value health based on mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Time Frame: The EQ-5D-5L is administered at baseline, six months and one year.
Population: The protocol states that this endpoint would be addressed if and only if the primary endpoint supports the primary hypothesis, therefore data is not reported.
Arm/Group | Sorafenib Alone | SBRT Followed by Sorafenib
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Overall Survival by Sex
Description: NIH-required analysis. An event for overall survival (OS) is death due to any cause. Survival time is defined as time from randomization to the date of death or last known follow-up (censored). Rates are estimated by the Kaplan-Meier method. Analysis was to occur after 153 deaths were reported.
Time Frame: as for outcome 1
Population: Eligible participants. Data were stratified by sex.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Sorafenib Alone | SBRT Followed by Sorafenib
Number analyzed (Participants) | 92 | 85
months
  Female: number analyzed (Participants) | 10 | 17
  Female | 13.80 [4.21 to 31.80] | 10.68 [7.07 to 15.29]
  Male: number analyzed (Participants) | 82 | 68
  Male | 12.30 [10.62 to 14.30] | 17.08 [13.35 to 21.53]

9. Other Pre Specified Outcome: Overall Survival by Ethnicity
Description: as for outcome 8
Time Frame: as for outcome 1
Population: Eligible participants. Data were stratified by ethnicity.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Sorafenib Alone | SBRT Followed by Sorafenib
Number analyzed (Participants) | 92 | 85
months
  Hispanic or Latino: number analyzed (Participants) | 6 | 2
  Hispanic or Latino | 10.48 [4.70 to 13.25] | 17.80 [6.81 to 28.80]
  Not Hispanic or Latino: number analyzed (Participants) | 54 | 47
  Not Hispanic or Latino | 12.11 [8.63 to 17.28] | 15.29 [10.98 to 17.95]
  Unknown or Not Reported: number analyzed (Participants) | 32 | 36
  Unknown or Not Reported | 13.16 [9.14 to 17.60] | 15.85 [11.31 to 21.24]

10. Other Pre Specified Outcome: Overall Survival by Race
Description: as for outcome 8
Time Frame: as for outcome 1
Population: Eligible participants. Data were stratified by race.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Sorafenib Alone | SBRT Followed by Sorafenib
Number analyzed (Participants) | 92 | 85
months
  American Indian or Alaska Native: number analyzed (Participants) | 1 | 0
  American Indian or Alaska Native | 10.65 [NA to NA] — Lower and upper confidence bounds cannot be estimated because the analysis includes only one subject. |
  Asian: number analyzed (Participants) | 23 | 18
  Asian | 12.30 [4.60 to 17.60] | 18.23 [11.31 to 26.76]
  Native Hawaiian or Other Pacific Islander: number analyzed (Participants) | 0 | 1
  Native Hawaiian or Other Pacific Islander |  | 2.10 [NA to NA] — Lower and upper confidence bounds cannot be estimated because the analysis includes only one subject.
  Black or African American: number analyzed (Participants) | 5 | 3
  Black or African American | 7.35 [3.55 to NA] — Upper confidence bound could not be estimated because the upper confidence limit for survival did not cross 50% | 20.35 [10.94 to 29.76]
  White: number analyzed (Participants) | 58 | 59
  White | 12.03 [10.32 to 14.70] | 14.70 [11.21 to 20.28]
  Unknown or not reported: number analyzed (Participants) | 5 | 4
  Unknown or not reported | 22.88 [13.08 to NA] — Upper confidence bound could not be estimated because the upper confidence limit for survival did not cross 50% | 11.94 [5.34 to 39.22]

ADVERSE EVENTS:
Time Frame: From randomization to last follow-up: weekly during SBRT, after SBRT and before starting sorafenib, monthly during sorafenib, and overall from study entry: every 3 months for 2 years, then every 6 months. Maximum follow-up at time of analysis was 7.6 years.
Description: All-cause mortality was assessed in eligible participants. Adverse events were assessed in eligible participants who started protocol treatment, and were assessed for adverse events.
Arm/Group | Sorafenib Alone | SBRT Followed by Sorafenib
All-Cause Mortality (participants affected / at risk) | 80/92 | 73/85
Serious Adverse Events (participants affected / at risk) | 20/88 | 19/83
Other Adverse Events (participants affected / at risk) | 88/88 | 83/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib Alone (N=88) | SBRT Followed by Sorafenib (N=83)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Ascites (Gastrointestinal disorders) | 0 | 2
Duodenal perforation (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 3
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1
Death NOS (General disorders) | 1 | 0
Flu like symptoms (General disorders) | 2 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 4 | 1
Hepatic hemorrhage (Hepatobiliary disorders) | 1 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 1
Bone infection (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 2
Lung infection (Infections and infestations) | 0 | 1
Peritoneal infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 2 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 1
Visceral arterial ischemia (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib Alone (N=88) | SBRT Followed by Sorafenib (N=83)
Anemia (Blood and lymphatic system disorders) | 25 | 44
Abdominal distension (Gastrointestinal disorders) | 10 | 3
Abdominal pain (Gastrointestinal disorders) | 29 | 28
Ascites (Gastrointestinal disorders) | 7 | 11
Bloating (Gastrointestinal disorders) | 2 | 8
Constipation (Gastrointestinal disorders) | 21 | 16
Diarrhea (Gastrointestinal disorders) | 43 | 38
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 15 | 19
Gastrointestinal pain (Gastrointestinal disorders) | 5 | 5
Mucositis oral (Gastrointestinal disorders) | 7 | 6
Nausea (Gastrointestinal disorders) | 28 | 37
Vomiting (Gastrointestinal disorders) | 9 | 18
Edema limbs (General disorders) | 12 | 14
Fatigue (General disorders) | 55 | 54
Fever (General disorders) | 7 | 3
General disorders and administration site conditions - Other, specify (General disorders) | 10 | 14
Pain (General disorders) | 6 | 8
Infections and infestations - Other, specify (Infections and infestations) | 5 | 4
Activated partial thromboplastin time prolonged (Investigations) | 2 | 5
Alanine aminotransferase increased (Investigations) | 31 | 40
Alkaline phosphatase increased (Investigations) | 14 | 22
Aspartate aminotransferase increased (Investigations) | 45 | 41
Blood bilirubin increased (Investigations) | 49 | 54
Creatinine increased (Investigations) | 8 | 4
INR increased (Investigations) | 8 | 19
Investigations - Other, specify (Investigations) | 17 | 24
Lymphocyte count decreased (Investigations) | 8 | 18
Neutrophil count decreased (Investigations) | 16 | 19
Platelet count decreased (Investigations) | 49 | 63
Weight loss (Investigations) | 22 | 19
White blood cell decreased (Investigations) | 16 | 38
Anorexia (Metabolism and nutrition disorders) | 39 | 34
Hyperglycemia (Metabolism and nutrition disorders) | 10 | 17
Hypoalbuminemia (Metabolism and nutrition disorders) | 40 | 41
Hypocalcemia (Metabolism and nutrition disorders) | 20 | 18
Hypokalemia (Metabolism and nutrition disorders) | 4 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 17 | 17
Hyponatremia (Metabolism and nutrition disorders) | 28 | 16
Hypophosphatemia (Metabolism and nutrition disorders) | 32 | 32
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 15 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 | 3
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 14 | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 3
Dysgeusia (Nervous system disorders) | 4 | 5
Headache (Nervous system disorders) | 12 | 7
Nervous system disorders - Other, specify (Nervous system disorders) | 5 | 1
Insomnia (Psychiatric disorders) | 13 | 7
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 12
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 8
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 28 | 21
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 9
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 21 | 17
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 23 | 14
Hypertension (Vascular disorders) | 24 | 20

LIMITATIONS AND CAVEATS:
The trial closed to accrual in March 2021 at 193 of 292 planned patients due to a change in the systemic standard of care for this disease, from sorafenib to atezolizumab and bevacizumab. As the original number of OS events (238) couldn't be met, the statistical analysis plan (SAP) was revised to report the study using available patients, with data through 7/1/2022. The changes were done by a statistician independent from the trial in accordance with the NCI Policy for Major Design Amendments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT01730937/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT01730937/ICF_001.pdf